CLINICAL TRIAL: NCT07296653
Title: Efficacy of Prolotherapy in Acupoints in Chronic Non-specific Low Back Pain (cLBP) - A Randomized Control Trial
Brief Title: Prolotherapy in Acupoints in Chronic Non-specific Low Back Pain (cLBP)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Konstantinos Kalimeris, Associate Professor of Anesthesiology, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 621, 12.09.2025
Record Dates: First submitted 2025-11-16; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Chronic Non-specific Low Back Pain
Keywords: prolotherapy; acupoints; dextrose; low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Glucose; Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine (Sham Comparator): Infiltration of back acupoints with lidocaine 1%
  Interventions: Drug: Lidocaine 1% infiltration
- Dextrose and lidocaine (Active Comparator): Infiltration of back acupoints with dextrose 15% and lidocaine 1%
  Interventions: Drug: Dextrose 15% and lidocaine 1% infiltration

INTERVENTIONS:
Drug: Dextrose 15% and lidocaine 1% infiltration — Infiltration of back acupoints
  Arms: Dextrose and lidocaine
Drug: Lidocaine 1% infiltration — Infiltration of dextrose and lidocaine in back acupoints
  Arms: Lidocaine

SUMMARY:
Chronic non-specific low back pain (CNSLBP) is among the most prevalent causes of disability on the planet, which often proves to be refractory to conventional pharmacological, interventional, and rehabilitation approaches. Although acupuncture has also shown analgesic effectiveness, its variability and reliance on practitioner skill limit its universal introduction into Western medical practice. Prolotherapy, an emerging regenerative injection treatment with hypertonic dextrose solutions, has been of potential benefit in managing musculoskeletal pain by triggering tissue repair and controlling neurogenic inflammation. Interestingly, several acupuncture points correspond to neuroanatomically relevant sites.

This single-blind randomized controlled trial aims to ascertain whether combinational prolotherapy with dextrose 15% and lidocaine 1% is superior to lidocaine 1% in patients with CNSLBP. Sixty patients will be allocated randomly into two equal-sized groups and receive a maximum of 15 ultrasound-guided injections into standardized acupoints of the lumbar area (BL23, BL25, BL31, BL54, GV3, GV4, and Ashi points) during three treatment sessions. Outcomes will be evaluated using the Numeric Rating Scale (NRS), the Oswestry Disability Index (ODI), the TUG (Timed Up and Go) test, the BPI (Brief Pain Inventory) scale, the Rolland-Morris Low Back Pain Disability Questionnaire and the Global Impression of Pain Questionnaire at baseline, and at 15, 30, and 90 days post-treatment.

Outcomes should clarify whether dextrose-enhanced prolotherapy provides improved analgesia and functional return in comparison with local anesthetic injection alone. This study can present an uncomplicated, low-cost, and integrative regimen for CNSLBP with significant clinical and socioeconomic implications.

DETAILED DESCRIPTION:
Background and Rationale Chronic non-specific low back pain (CNSLBP) is among the most prevalent and disabling musculoskeletal conditions in the world, with approximately 60-80% of individuals developing it at some point during their lifetime. Unlike specific etiologies for back pain, e.g., fracture, infection, or radiculopathy, CNSLBP has no explicitly diagnosable pathological or structural cause. Yet, it often leads to chronic pain, functional disability, and reduced quality of life. The economic burden of CNSLBP extends beyond the patient, with high socioeconomic costs in healthcare consumption, lost productivity, and disability-related absenteeism. Despite extensive use of conventional treatments, e.g., pharmacologic treatments, physiotherapy, and interventions, most patients are only temporarily or partially relieved, indicating an urgent requirement for an improved long-term management regimen.

Traditional Western medical interventions have a proclivity to address inflammatory or structural causes, and conventional pharmacotherapy generally provides transient symptom relief of limited duration. NSAIDs, muscle relaxants, and opioids can abate acute symptoms but are side-affected and of little long-term efficacy. Similarly, interventional therapies, i.e., epidural steroid injection or radiofrequency ablation, may be targeted at specific anatomical structures but do not address the multifactorial causation of CNSLBP and resultant recurrence or chronicity of pain. Complementary treatments, e.g., exercise, cognitive behavior therapy, and acupuncture, are inconsistently effective, and integration into mainstream clinical practice is frequently disrupted by complexity, cost, or the need for special training.

Prolotherapy, or proliferative therapy, is a new regenerative therapy for chronic musculoskeletal pain. Hypertonic dextrose solution injections near ligaments, tendons, and periarticular tissue is postulated to enhance local repair of tissue, collagen production, and modulation of neurogenic inflammation in dextrose prolotherapy. Targeted injections, based on recent studies, reduce pain and improve function, particularly in chronic low back pain that is resistant to conventional treatment. Of note, many of the anatomic sites treated with prolotherapy are also points for acupuncture, which have been shown to influence neurovascular physiology, endogenous opioid release, and pain modulatory systems. This overlap provides a unique venue for the convergence of the mechanistic benefits of both interventions.

Despite encouraging early findings, few studies have assessed the efficacy of prolotherapy in patients with CNSLBP systematically. There is not much evidence to support prolotherapy; that's why it has not been widely practiced. The treatment site is also non-uniform. This is why we would like to conduct this study, as a way of finding out whether the protocol of prolotherapy to and from universally recognized lumbar acupoints can provide clinically meaningful reductions in pain severity and improvement in functional capability, and thus address a highly important unmet need in the treatment of chronic low back pain.

Study Objectives and Hypotheses The primary study objective is to determine the clinical effectiveness of combinational prolotherapy injectate delivered to standardized acupuncture points for the management of adults with chronic non-specific low back pain (CNSLBP). Specifically, we wish to determine whether the intervention has a significant impact on reducing pain intensity and enhancing functional ability compared with the use of local anesthetic injections alone. By stimulating acupoints that correspond to the lumbar region, this approach is designed to combine regenerative, neuromodulatory, and analgesic mechanisms that may offer a more comprehensive solution for those who remain symptomatic despite conventional therapies.

Secondary objectives are to assess the impact of the intervention on quality of life, patient-reported disability, and global physical performance, as measured by validated instruments of pain and mobility assessment, such as:

* the Oswestry Disability Index (ODI)
* the Numeric Rating Scale (NRS)
* the BPI (Brief Pain Inventory) scale
* the TUG (Timed UP and Go Functional Low Back Pain Test)
* the Roland-Morris (Low Back Pain disability questionnaire)
* the GIC (Global Impression of Change) Scale Safety and tolerability will be tracked by reporting of injection-related adverse events. We also wish to ascertain whether treatment at specific acupoints is linked with differential effects, thereby providing initial data concerning point-specific efficacy.

The study aims to test the following hypotheses:

1. Primary Hypothesis: The patients treated with prolotherapy at standardized lumbar acupuncture points will experience a clinically appreciable reduction in pain intensity and improved functional outcomes compared to those treated with local anesthetic injections alone.
2. Secondary Hypotheses:

   * Patient-reported disability and quality of life scores will be improved by the intervention.
   * The treatment will be safe and well-tolerated with minimal adverse effects. By setting out these well-defined objectives and hypotheses, this study seeks to provide robust evidence on the effectiveness and safety of combinational prolotherapy for CNSLBP, a highly needed area in the management of chronic musculoskeletal pain.

Study Design This study is a prospective, single-blind, randomized controlled trial (RCT) with the aim of determining the effectiveness of combinational prolotherapy in patients with chronic non-specific low back pain (CNSLBP). 60 adult participants will be enrolled and randomized in a 1:1 ratio to the intervention group ("Prolo Group") or active control group ("Lido Group"). Randomization will be achieved using computer-generated sequences to allow allocation concealment, minimizing selection bias. Participants will be blinded to group assignments, but clinicians who will be giving the injections will not be blinded due to the nature of the intervention. This single-blind design balances methodological rigor and practicality.

The Prolo Group will receive injections of hypertonic dextrose solution (15% D-glucose) with 1% lidocaine, injected into up to 15 lumbar acupuncture points per session. The Lido Group will receive injections of 1% lidocaine, the same procedure, as an active comparator to control for mechanical needle and local anesthetic effects. For each injection, a 23G, 25 mm needle with 1 mL of solution will be used. Ultrasound guidance will be employed to accurately identify anatomical targets, while palpation will be used to locate tender or Ashi points consistent with the standardized protocol.

Treatment will be administered in three sessions: one baseline session, a second session at two weeks, and a third session at four weeks. Follow-up visits will occur at 15, 30, and 90 days after the last injection to determine both short- and medium-term effects. The design provides the opportunity to observe cumulative effects, temporal characteristics of pain relief, and functional change.

Participants The research will recruit 60 adult patients with chronic non-specific low back pain (CNSLBP) as a defined condition of persistent lumbar pain greater than three months' duration without apparent structural, inflammatory, neoplastic, or neurological pathology. Recruitment will be by referral from outpatient pain clinics and primary care physicians and through targeted advertisements in health centers, providing a representative sample akin to real-life patient populations.

Baseline measurements will include demographic data, medical history, and initial pain and disability scores. Tender points will be systematically mapped consistent with the uniform acupuncture protocol, so that identical targeting is achieved on injection. Participants will also be provided advice on permissible concomitant treatments, and limits will be imposed on the initiation of new interventional treatments or alteration of current analgesic therapy during the study.

This clearly delineated participant population ensures that the research examines combinational prolotherapy effects in a representative CNSLBP cohort with rigorous safety protocols. Strict inclusion and exclusion criteria and methodical baseline assessments will allow for accurate measurement of treatment outcomes and replicability of the results.

Intervention Procedures The intervention protocol in this study is to determine the effects of combinational prolotherapy injected at standardized lumbar acupuncture points, consisting of regenerative and analgesic processes. Two groups will be randomized for participants: the Prolo Group, in which the participants will be injected with combinational prolotherapy with hypertonic dextrose and lidocaine, and the Lido Group, in which participants will be injected with local anesthetic injections alone. The purpose is to see whether the administration of dextrose provides additional clinical value beyond mechanical needle effects and local anesthetic action.

Injection Materials and Preparation

* Prolo Group: All participants will receive 15% dextrose (D-glucose) with 1% lidocaine.
* Lido Group: All participants will receive 1% lidocaine alone. Solutions will be prepared fresh in a sterile environment immediately before each session. All injections are 1 mL per location.

Point Selection Injection sites are standardized based on a modified acupoint protocol for the most widely utilized lumbar points associated with chronic low back pain. These include BL23 (Shenshu), BL25 (Dachangshu), BL31 (Shangliao), BL54 (Zhibian), GV3 (Yaoyangguan), GV4 (Mingmen), and patient-specific Ashi points accessed by palpation.

Procedural Steps

1. Localization: Points will be found before injection by means of ultrasound and palpation.
2. Injection Technique: The needle will be inserted perpendicularly into the target site, following skin antisepsis, and the solution to be administered will be injected slowly over the course of a few seconds. Gently used tissue manipulation can facilitate diffusion.
3. Session Schedule: There will be three sessions administered to the subjects: a baseline injection as the initial session, the second session in two weeks' time, and the third session four weeks later. The sessions should last approximately 25-30 minutes.
4. Post-procedure Care: The participants will be observed for 15-20 minutes post-injection for side effects. Routine post-procedure care, like activity modification and watchful waiting for late reactions, will be provided.

Measurements:

Change in pain, measured through:

* the BPI (Brief Pain Inventory) scale: Baseline evaluation and d90 following the end of the infiltrations (injection sessions). Patients are asked to rate their pain on a 0 (no pain) to 10 (worst possible pain) scale.
* the Numeric Rating Scale (NRS): 15 minutes after every infiltration (1st, 2nd and 3rd), d15 and d30 after the 3rd infiltration. This measure provides a valid, sensitive, patient-centered measure of pain experience with the ability to detect clinically significant change over time.

Functional Disability (activity limitations due to low back pain), measured through:

* the Oswestry Disability Index (ODI): Baseline evaluation, d15, d30 and d90 after 3rd infiltration. It is a ten-item self-administered questionnaire covering personal care, lifting, walking, and social life, scored in percentages. The higher score indicates more disability.
* the TUG (Timed UP and Go Functional Low Back Pain Test): Baseline evaluation, 15 minutes before and after 1st Infiltration and d15, d30, and d90 after 3rd infiltration
* Pain reduction, duration of analgesia, and optimism at 24h after the end of the first session. Pain reduction after the first session will be analyzed as a predictor of the pain improvement 1 month after the end of the 3 sessions.
* the Roland-Morris (Low Back Pain disability questionnaire): Baseline evaluation, d15 and d90 after 3rd infiltration
* the GIC (Global Impression of Change) Scale: d90 after 3rd Infiltration. Participants will provide a rating of overall change on a 7-point Likert scale, indicating subjective assessment of the effectiveness of the treatment.

Safety and Tolerability Adverse events will be recorded routinely at all sessions and follow-up. Minor common reactions should be short-lasting injection-site pain or bruising. Serious adverse events, though unlikely given the minimally invasive procedure, will be reported immediately and reviewed by the study's safety monitoring committee.

Assessment Schedule

* Baseline: Demographics, medical history, and tender points and initial questionnaires.
* During Intervention: Pre-injection NRS scores at each session (weeks 0, 2, and 4) and follow-up for immediate adverse events.
* Follow-Up: Global reassessment at 15, 30, and 90 days post-last injection, encompassing the aforementioned questionnaires and scales.

Contact and questions 24h after the first intervention.

This multi-level evaluation strategy ensures robust analysis of short- and medium-term impact, providing extensive insight into the intervention's clinical effect and safety profile. The study captures both objective and subjective treatment response with the combination of established quantitative measures and patient-reported outcomes.

Statistical Analysis Statistical analysis design is attracted to critically evaluate the safety and efficacy of combinational prolotherapy in treating chronic non-specific low back pain (CNSLBP), with proper regard to transparency, reproducibility, and concomitance with standard clinical research methods.

Sample Size Calculation Sample size was estimated based on previous studies on prolotherapy and injection therapy for CNSLBP (Maniquis-Smigel 2017; Sirh et al. 2022). To adress potential dropouts and keep enough power, the study will include 60 participants divided evenly between the Prolo Group (dextrose + lidocaine) and the Lido Group (lidocaine alone).

The trial shall be run for a duration of about 18-24 months with separate phases of recruitment, intervention, follow-up, and analysis of data. Time has been factored in for anticipated recruitment rates, retention among the participants, and the sequential nature of the intervention protocol.

Possible Benefits Participants of the study can anticipate various benefits in terms of clinical outcomes. The most anticipated benefit is the reduction in pain severity as assessed with the Numeric Rating Scale (NRS), and this can enhance daily functioning and quality of life. Secondary benefits could include enhanced mobility, reduced disability as measured by the Oswestry Disability Index (ODI), and improvements in physical and psychosocial status. The targeted injections also have the capability to produce localized effects via modulation of peripheral nerve sensitization, tissue repair, and enhancement of microcirculation within the affected tissue. Furthermore, the study will create standardized protocols for combinational prolotherapy at common acupuncture points, which would be applicable to future clinical treatments and result in evidence-based practices for treating chronic low back pain. Participants will also profit from structured education, exercise teaching, and lifestyle counseling, part of the study, which will support extended self-management practice.

Potential Risks This therapy does not entail any risks at all, being non-systemic in practice and executed under aseptic conditions. Slight, usual side effects are brief discomfort, slight bruising, or soreness at the injection sites. Some may also experience temporary local swelling or erythema. Use of a mixture of dextrose and lidocaine is intended to reduce discomfort during the injections. Serious complications, such as infection, bleeding, or nerve injury, are highly unlikely due to the superficiality of the injections and adherence to strict aseptic protocol.

Ethical Considerations Participating individuals shall be completely informed about the potential risks and benefits prior to providing their written consent. The study shall adhere to strict ethical principles, including ongoing safety monitoring, participants' right to withdraw at any time, and provision for rescue therapies in the event of an inadequate response.

In summary, the potential benefits of relief from pain, enhanced functioning, and the gain in scientific information considerably outweigh the minimal and manageable risks of the intervention and hence justify the ethical justification for conducting this study.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) up to 45 kg/m2
* Diagnoses corresponding to >1 of the following ICD-10 (International Classification of Diseases):

  1. M51.3 Degeneration of intervertebral discs
  2. M54.5 Low back pain
  3. M54.8 Other forms of back pain
  4. M54.9 Various forms of back pain
  5. S33.5 Sprain of the lumbar spine
  6. S33.6 Sprain of sacroiliac joint
  7. S33.7 Sprain of other and various parts of lumbar spine and pelvis
* Diagnosis of chronic nonspecific low back pain: Chronic nonspecific low back pain refers to pain in the lower back with or without radiation to the lower extremities, lasting for more than 3 months and not attributable to a specific anatomical structure or pathology on imaging, for example generalized degenerative changes, but no pathological findings (such as spinal stenosis or disorders of the sagittal/coronal architecture or intervertebral foramen stenosis) with neurological deficits and no symptoms specific to the predominant pathology.
* Numerical Rating Scale (NRS) > 3/10 for at least 3 months prior to the study
* Positive response to >1 muscle strength assessment tests in chronic low back pain A. prone plank bridge test (PBT) B. side bridge test (SBT) C. supine bridge test (SUBT) D. Range of Motion (ROM) E. Back Performance Scale (BPS) F. Straight leg raise test (SLR)
* Pain, inability to walk, and stiffness in the lumbar spine, persisting for at least three months prior to the study.
* Radiological imaging tests such as MRI or CT and, in cases of clinical suspicion (where appropriate), X-rays with dynamic flexion/extension or whole spine X-rays.
* Signing of written consent prior to the injection of pharmaceutical agents.

Exclusion Criteria:

* Any infection of the skin of the lumbar spine area, such as cellulitis, or periarticular or intra-articular infection or spondylodiscitis during the last 3 months
* History of periarticular or intra-articular injection in the LMS with corticosteroids, local anesthetic, hyaluronic acid, radiofrequency application, electroacupuncture, or prolotherapy within the last three months.
* Previous surgery (e.g., spinal fusion) in the LMS
* Oral corticosteroids for low back pain or uncontrolled opioids
* History of the following diseases:

  1. connective tissue disease affecting the intervertebral spaces
  2. insulin-dependent diabetes mellitus without adequate control
  3. acute lumbosacral radiculopathy or peripheral neuropathy
  4. neurological/psychiatric disease
  5. history of malignancy in the area or any other active malignancy in the body
  6. Bleeding disorder
  7. Trauma during the previous three months without imaging investigation
  8. Systemic diseases such as rheumatic diseases
  9. Known abdominal aortic aneurysm
* Pregnancy (based on history)
* History of allergy to local anesthetics
* Needle phobia
* Inability to communicate adequately, severe hearing loss, language problems, dementia
* Inability to guarantee transportation to the hospital for treatments/follow-up examinations

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Pain severity score 15 days after completion of the intervention | 15 days after completion of infiltrations of first participant until 15 days after completion of infiltration of the last participant.
  Pain severity score from the short Brief Pain Inventory (BPI) form, 15 days after completion of the infiltrations.
  Minimum value: 0 and Maximum value: 10 Higher scores correspond to worse outcome - i.e. greater pain severity or greater interference with functioning.

SECONDARY OUTCOMES:
Pain severity score at 90 days after completion of the therapy | From 90 days after completion of the infiltrations of the first participant until 1 month after completion of infiltrations of the last participant. Just before the first infiltration a baseline measurement will be also made.
  Pain severity score from BPI short form 90 days after completion of the infiltrations.
Oswestry disability index (ODI) at baseline, 15, 30 and 90 days after completion of therapy | Before first infiltration of the first participant up to 3 months after completion of the therapy of the last one.
  Oswestry scale score
Short term changes after the first infiltration | 24 hours (Day 1) after first infiltration of the first participant until 24 hours after first infiltration of the last participant.
  Pain decrease, duration of analgesia and optimism at 24 hours (Day 1) after completion of the first session. Pain reduction after the first session will be analyzed as prognostic factor for the pain improvement.
TUG (timed up and go) test | Just before the first infiltration until 3 months after completion of the therapy of the last participant
  TUG test in seconds at baseline, 15 minutes before and after 1st Infiltration and Day 15, Day 30, and Day 90 after the 3rd infiltration
Global impression of change | From one month after completion of therapy of the first participant until 3 months after completion of therapy of the last participant.
  Global impression of change 90 days after completion of the therapy
Roland-Morris Low Back Pain disability questionnaire | Baseline evaluation, Day 15 and Day 90 after the 3rd infiltration
  Baseline evaluation, Day 15 and Day 90 after the 3rd infiltration
Pain intensity score after completion of the interventions programmed | Day 1, Day 7, Day 15, Day 30, Day 90 after the infiltrations
  Pain severity score from the Numeric Rating Scale (0-10) used to quantify pain intensity (0=no pain, 10=worst pain imaginable)

OTHER OUTCOMES:
Subanalyses of the scales measured | Time frames are pre-determined as stated from the above mentioned scales: DAY 1, DAY 15, DAY 30, (immediately after the interventions), DAY 90 after the first infiltration
  Subanalyses of questions from the above mentioned scales (BPI + Oswestry Disability Index + Rolland + TUG + ΝRS + Global Impression of Change) eg. usage of analgesics, changes in life attitudes, changes in movement/work/food habits, undergoing other parallel treatments or hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Kalimeris, Assoc Prof of Anesthesiology, Study Chair — National and Kapodistrian University of Athens; Theodosios Saranteas, Professor of Anesthesiology, Study Chair — National and Kapodistrian University of Athens; Lampis Stavrinou, Assist Prof of Neurosurgery, Study Chair — National and Kapodistrian University of Athens
Locations (1):
- University General Hospital of Athens "Attikon" - National and Kapodistrian University of Athens Medical School, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes
Responses to Questionnaires (NRS, Rolland-Morris, Oswestry, GIC, TUG)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: They will be available from the end of the recording of the response of the last patient to the infiltrations and for 5 years thereafter.
Access Criteria: Researchers that would have come in contact with our team firstly and that shall be able to prove that they will use the data solely for research purposes and not for commercial use.
URL: https://attikonhospital.gov.gr/

REFERENCES:
- [Background] Shumway-Cook A, Brauer S, Woollacott M. Predicting the probability for falls in community-dwelling older adults using the Timed Up & Go Test. Phys Ther. 2000 Sep;80(9):896-903. PMID 10960937
- [Background] Caserta F, Stanley HE, Eldred WD, Daccord G, Hausman RE, Nittmann J. Physical mechanisms underlying neurite outgrowth: A quantitative analysis of neuronal shape. Phys Rev Lett. 1990 Jan 1;64(1):95-98. doi: 10.1103/PhysRevLett.64.95. No abstract available. PMID 10041282
- [Background] Walton J. Educating the doctor: basic medical education. Br Med J (Clin Res Ed). 1985 Jun 8;290(6483):1719-22. doi: 10.1136/bmj.290.6483.1719. No abstract available. PMID 3924230
- [Background] Han SP, Han JS. Acupuncture and Related Techniques for Pain Relief and Treatment of Heroin Addiction: Mechanisms and Clinical Application. Med Acupunct. 2020 Dec 1;32(6):403-404. doi: 10.1089/acu.2020.1485. Epub 2020 Dec 16. PMID 33362900
- [Background] Koldas Dogan S, Sonel Tur B, Kurtais Y, Atay MB. Comparison of three different approaches in the treatment of chronic low back pain. Clin Rheumatol. 2008 Jul;27(7):873-81. doi: 10.1007/s10067-007-0815-7. Epub 2008 Jan 11. PMID 18188660
- [Background] Last AR, Hulbert K. Chronic low back pain: evaluation and management. Am Fam Physician. 2009 Jun 15;79(12):1067-74. PMID 19530637
- [Background] Fan Z, Dou B, Wang J, Wu Y, Du S, Li J, Yao K, Li Y, Wang S, Gong Y, Guo Y, Xu Z. Effects and mechanisms of acupuncture analgesia mediated by afferent nerves in acupoint microenvironments. Front Neurosci. 2024 Feb 7;17:1239839. doi: 10.3389/fnins.2023.1239839. eCollection 2023. PMID 38384495
- [Background] Andersson GB. Epidemiological features of chronic low-back pain. Lancet. 1999 Aug 14;354(9178):581-5. doi: 10.1016/S0140-6736(99)01312-4. PMID 10470716
- [Background] Mauck MC, Aylward AF, Barton CE, Birckhead B, Carey T, Dalton DM, Fields AJ, Fritz J, Hassett AL, Hoffmeyer A, Jones SB, McLean SA, Mehling WE, O'Neill CW, Schneider MJ, Williams DA, Zheng P, Wasan AD. Evidence-based interventions to treat chronic low back pain: treatment selection for a personalized medicine approach. Pain Rep. 2022 Sep 30;7(5):e1019. doi: 10.1097/PR9.0000000000001019. eCollection 2022 Sep-Oct. PMID 36203645
- [Background] Hayden JA, Ellis J, Ogilvie R, Malmivaara A, van Tulder MW. Exercise therapy for chronic low back pain. Cochrane Database Syst Rev. 2021 Sep 28;9(9):CD009790. doi: 10.1002/14651858.CD009790.pub2. PMID 34580864
- [Background] Edwards RR, Schreiber KL, Dworkin RH, Turk DC, Baron R, Freeman R, Jensen TS, Latremoliere A, Markman JD, Rice ASC, Rowbotham M, Staud R, Tate S, Woolf CJ, Andrews NA, Carr DB, Colloca L, Cosma-Roman D, Cowan P, Diatchenko L, Farrar J, Gewandter JS, Gilron I, Kerns RD, Marchand S, Niebler G, Patel KV, Simon LS, Tockarshewsky T, Vanhove GF, Vardeh D, Walco GA, Wasan AD, Wesselmann U. Optimizing and Accelerating the Development of Precision Pain Treatments for Chronic Pain: IMMPACT Review and Recommendations. J Pain. 2023 Feb;24(2):204-225. doi: 10.1016/j.jpain.2022.08.010. Epub 2022 Oct 2. PMID 36198371
- [Background] Strudwick MW, Hinks RC, Choy ST. Point injection as an alternative acupuncture technique--an exploratory study of responses in healthy subjects. Acupunct Med. 2007 Dec;25(4):166-74. doi: 10.1136/aim.25.4.166. PMID 18160927
- [Background] Giordano L, Murrell WD, Maffulli N. Prolotherapy for chronic low back pain: a review of literature. Br Med Bull. 2021 Jun 10;138(1):96-111. doi: 10.1093/bmb/ldab004. PMID 33884404
- [Background] Knezevic NN, Mandalia S, Raasch J, Knezevic I, Candido KD. Treatment of chronic low back pain - new approaches on the horizon. J Pain Res. 2017 May 10;10:1111-1123. doi: 10.2147/JPR.S132769. eCollection 2017. PMID 28546769
- [Background] Sirh SJ, Sirh SW, Mun HY, Sirh HM. Importance of quadratus lumborum muscle trigger point injection and prolotherapy technique for lower back and buttock pain. Front Pain Res (Lausanne). 2022 Nov 22;3:997645. doi: 10.3389/fpain.2022.997645. eCollection 2022. PMID 36483943
- [Background] Singh S, Patel AA, Singh JR. Intervertebral Disc Degeneration: The Role and Evidence for Non-Stem-Cell-Based Regenerative Therapies. Int J Spine Surg. 2021 Apr;15(s1):54-67. doi: 10.14444/8055. Epub 2021 Apr 19. PMID 34376496
- [Background] Hauser RA, Matias D, Woznica D, Rawlings B, Woldin BA. Lumbar instability as an etiology of low back pain and its treatment by prolotherapy: A review. J Back Musculoskelet Rehabil. 2022;35(4):701-712. doi: 10.3233/BMR-210097. PMID 34957989
- [Background] Chen CPC, Suputtitada A. Prolotherapy at Multifidus Muscle versus Mechanical Needling and Sterile Water Injection in Lumbar Spinal Stenosis. J Pain Res. 2023 Jul 18;16:2477-2486. doi: 10.2147/JPR.S417444. eCollection 2023. PMID 37483410
- [Background] Dagenais S, Yelland MJ, Del Mar C, Schoene ML. Prolotherapy injections for chronic low-back pain. Cochrane Database Syst Rev. 2007 Apr 18;2007(2):CD004059. doi: 10.1002/14651858.CD004059.pub3. PMID 17443537
- [Background] Wang F, Cheung CW, Wong SSC. Regenerative medicine for the treatment of chronic low back pain: a narrative review. J Int Med Res. 2023 Feb;51(2):3000605231155777. doi: 10.1177/03000605231155777. PMID 36802994
- [Background] Maniquis-Smigel L, Dean Reeves K, Jeffrey Rosen H, Lyftogt J, Graham-Coleman C, Cheng AL, Rabago D. Short Term Analgesic Effects of 5% Dextrose Epidural Injections for Chronic Low Back Pain: A Randomized Controlled Trial. Anesth Pain Med. 2016 Dec 6;7(1):e42550. doi: 10.5812/aapm.42550. eCollection 2017 Feb. PMID 28920043
- [Background] Furlan AD, Yazdi F, Tsertsvadze A, Gross A, Van Tulder M, Santaguida L, Gagnier J, Ammendolia C, Dryden T, Doucette S, Skidmore B, Daniel R, Ostermann T, Tsouros S. A systematic review and meta-analysis of efficacy, cost-effectiveness, and safety of selected complementary and alternative medicine for neck and low-back pain. Evid Based Complement Alternat Med. 2012;2012:953139. doi: 10.1155/2012/953139. Epub 2011 Nov 24. PMID 22203884
- [Background] Hauser RA, Lackner JB, Steilen-Matias D, Harris DK. A Systematic Review of Dextrose Prolotherapy for Chronic Musculoskeletal Pain. Clin Med Insights Arthritis Musculoskelet Disord. 2016 Jul 7;9:139-59. doi: 10.4137/CMAMD.S39160. eCollection 2016. PMID 27429562
- [Background] Acupoint injection for nonspecific chronic low back pain: A protocol of systematic review: Erratum. Medicine (Baltimore). 2019 Nov;98(45):e18084. doi: 10.1097/MD.0000000000018084. No abstract available. PMID 31702688
- [Background] DeBar LL, Justice M, Avins AL, Cook A, Eng CM, Herman PM, Hsu C, Nielsen A, Pressman A, Stone KL, Teets RY, Wellman R. Acupuncture for chronic low back pain in older adults: Design and protocol for the BackInAction pragmatic clinical trial. Contemp Clin Trials. 2023 May;128:107166. doi: 10.1016/j.cct.2023.107166. Epub 2023 Mar 27. PMID 36990274
- [Background] Cherkin DC, Sherman KJ, Hogeboom CJ, Erro JH, Barlow WE, Deyo RA, Avins AL. Efficacy of acupuncture for chronic low back pain: protocol for a randomized controlled trial. Trials. 2008 Feb 28;9:10. doi: 10.1186/1745-6215-9-10. PMID 18307808
- [Background] Lai P, Cheng S, Chen X, Cheng F, Cheng J, Xin M, Zhu D, Li Z, Wu X, Zeng F. The Emotion Regulation of Acupuncture in Chronic Low Back Pain: A Clinical Neuroimaging Protocol. J Pain Res. 2024 Mar 1;17:817-825. doi: 10.2147/JPR.S450589. eCollection 2024. PMID 38444878
- [Background] Barber J, Lodo F, Nugent-Head A, Zeng X. Comparative Techniques of Acupuncture and Dry Needling Intersecting with Trigger Point Physiology and Diagnostics: A Cross-Discipline Narrative Review. Med Acupunct. 2023 Oct 1;35(5):220-229. doi: 10.1089/acu.2023.0031. Epub 2023 Oct 17. PMID 37900872
- [Background] Roland M, Fairbank J. The Roland-Morris Disability Questionnaire and the Oswestry Disability Questionnaire. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3115-24. doi: 10.1097/00007632-200012150-00006. No abstract available. PMID 11124727
- [Background] Borg-Stein J, Stein J. Trigger points and tender points: one and the same? Does injection treatment help? Rheum Dis Clin North Am. 1996 May;22(2):305-22. doi: 10.1016/s0889-857x(05)70274-x. PMID 8860801
- See also: Related Info — https://journalofprolotherapy.com/